CLINICAL TRIAL: NCT03282279
Title: Retrospective Analysis of the Incidence of Complications From Transvaginal Oocyte Retrieval (TVOR).
Acronym: TVOR
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 17/17
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2017-09

CONDITIONS: In Vitro Fertilization
Keywords: oocyte retrieval; surgical complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TVOR population: The data have been collected from the Humanitas Fertility Center' Department database (ART.it) from all transvaginal oocyte retrieval procedures performed between 1996 and October 2016.
  Interventions: Procedure: TVOR

INTERVENTIONS:
Procedure: TVOR — Ultrasound guided transvaginal oocyte retrieval (TVOR) in deep sedation for IVF.

SUMMARY:
The investigators retrospectively analysed the complication rate of ultrasound guided transvaginal oocyte retrieval (TVOR) from all the procedures performed between 1996 and October 2016 in a tertiary level university based fertility clinic.

DETAILED DESCRIPTION:
Ultrasound guided transvaginal oocyte retrieval (TVOR) is nowadays gold standard techniques to collect oocyte after ovulation induction in Assisted Reproductive techniques (ART). It is a very safe technique with infectious complications of any kind occurring in just 1% (Bennett et al.) of all procedures, vaginal bleeding in 0 to 1.3% of the procedures (Ludwig et al., Bodri et al., Aragona et al.) and vascular, gastrointestinal and genitourinary (Grynberg et al. and Catanzarite and al.), injuries being extremely rare (Bennett et al.). Case reports account also for rarer complications such as ovarian abscess formation (Kelada & Ghan and Sharp et al.) pseudoanerysm formation (Bozdag et al. and Jayakrishnan et al.), uroretroperitoneum (Fiori et al.).

The rational of thestudy is to provide the percentages of complication from TVOR of the Fertility Center of Humanitas Research Hospital, also considering the development in time of technologies and techniques in Assisted Reproduction. Another rational is inquire whether there is any risk factor for such complications in order to try to prevent them in future procedures. The investigators performed a retrospective observational study including all the transvaginal oocyte retrieval procedures performed between 1996 and October 2016.

The data have been collected from the Humanitas Fertility Center' Department database (ART.it). Because of the retrospective nature of this study, a specific informed consent was not necessary.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent ultrasound guided transvaginal oocyte retrieval during the study period

Exclusion Criteria:

* none

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patients that patients that underwent ultrasound guided transvaginal oocyte retrieval during the study period were including in the analysis.
  No case was excluded.
Sampling Method: Probability Sample
Enrollment: 23827 (Actual)
Dates: Start 1996-06-23 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
complications rate | 20 years
  number of oocyte retrieval complications reported / number of procedures

SECONDARY OUTCOMES:
hospitalisation rate | 20 years
  number of oocyte retrieval complications reported that required a admission to the hospital/ number of procedures

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cirillo, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan; Elena Zannoni, MD, Study Chair — Humanitas Research Hospital IRCCS, Rozzano-Milan; Paolo E Levi Setti, MD, Study Director — Humanitas Research Hospital IRCCS, Rozzano-Milan

REFERENCES:
- [Background] Bennett SJ, Waterstone JJ, Cheng WC, Parsons J. Complications of transvaginal ultrasound-directed follicle aspiration: a review of 2670 consecutive procedures. J Assist Reprod Genet. 1993 Jan;10(1):72-7. doi: 10.1007/BF01204444. PMID 8499683
- [Background] Ludwig AK, Glawatz M, Griesinger G, Diedrich K, Ludwig M. Perioperative and post-operative complications of transvaginal ultrasound-guided oocyte retrieval: prospective study of >1000 oocyte retrievals. Hum Reprod. 2006 Dec;21(12):3235-40. doi: 10.1093/humrep/del278. Epub 2006 Jul 27. PMID 16877373
- [Background] Bodri D, Guillen JJ, Polo A, Trullenque M, Esteve C, Coll O. Complications related to ovarian stimulation and oocyte retrieval in 4052 oocyte donor cycles. Reprod Biomed Online. 2008 Aug;17(2):237-43. doi: 10.1016/s1472-6483(10)60200-3. PMID 18681998
- [Background] Aragona C, Mohamed MA, Espinola MS, Linari A, Pecorini F, Micara G, Sbracia M. Clinical complications after transvaginal oocyte retrieval in 7,098 IVF cycles. Fertil Steril. 2011 Jan;95(1):293-4. doi: 10.1016/j.fertnstert.2010.07.1054. Epub 2010 Aug 21. PMID 20727520
- [Background] Grynberg M, Berwanger AL, Toledano M, Frydman R, Deffieux X, Fanchin R. Ureteral injury after transvaginal ultrasound-guided oocyte retrieval: a complication of in vitro fertilization-embryo transfer that may lurk undetected in women presenting with severe ovarian hyperstimulation syndrome. Fertil Steril. 2011 Oct;96(4):869-71. doi: 10.1016/j.fertnstert.2011.07.1094. Epub 2011 Aug 11. PMID 21839435
- [Background] Catanzarite T, Bernardi LA, Confino E, Kenton K. Ureteral Trauma During Transvaginal Ultrasound-Guided Oocyte Retrieval: A Case Report. Female Pelvic Med Reconstr Surg. 2015 Sep-Oct;21(5):e44-5. doi: 10.1097/SPV.0000000000000176. PMID 25900060
- [Background] Kelada E, Ghani R. Bilateral ovarian abscesses following transvaginal oocyte retrieval for IVF: a case report and review of literature. J Assist Reprod Genet. 2007 Apr;24(4):143-5. doi: 10.1007/s10815-006-9090-9. Epub 2007 Feb 16. PMID 17450435
- [Background] Sharpe K, Karovitch AJ, Claman P, Suh KN. Transvaginal oocyte retrieval for in vitro fertilization complicated by ovarian abscess during pregnancy. Fertil Steril. 2006 Jul;86(1):219.e11-3. doi: 10.1016/j.fertnstert.2005.12.045. Epub 2006 May 23. PMID 16716320
- [Background] Bozdag G, Basaran A, Cil B, Esinler I, Yarali H. An oocyte pick-up procedure complicated with pseudoaneurysm of the internal iliac artery. Fertil Steril. 2008 Nov;90(5):2004.e11-3. doi: 10.1016/j.fertnstert.2008.02.010. Epub 2008 Apr 18. PMID 18423457
- [Background] Jayakrishnan K, Raman VK, Vijayalakshmi VK, Baheti S, Nambiar D. Massive hematuria with hemodynamic instability--complication of oocyte retrieval. Fertil Steril. 2011 Jul;96(1):e22-4. doi: 10.1016/j.fertnstert.2011.04.046. Epub 2011 May 19. PMID 21600575
- [Background] Fiori O, Cornet D, Darai E, Antoine JM, Bazot M. Uro-retroperitoneum after ultrasound-guided transvaginal follicle puncture in an oocyte donor: a case report. Hum Reprod. 2006 Nov;21(11):2969-71. doi: 10.1093/humrep/del252. Epub 2006 Aug 29. PMID 16940321
- [Derived] Levi-Setti PE, Cirillo F, Scolaro V, Morenghi E, Heilbron F, Girardello D, Zannoni E, Patrizio P. Appraisal of clinical complications after 23,827 oocyte retrievals in a large assisted reproductive technology program. Fertil Steril. 2018 Jun;109(6):1038-1043.e1. doi: 10.1016/j.fertnstert.2018.02.002. Epub 2018 Jun 2. PMID 29871795